CLINICAL TRIAL: NCT03365024
Title: Computerized Cognitive Behavioral Treatment for Insomnia: Improving Rural Veteran Access to Evidence-Based Treatment to Reduce Suicide Risk
Brief Title: Computerized Cognitive Behavioral Treatment for Insomnia: Improving Rural Veteran Access to Evidence-Based Treatment to Reduce Suicide Risk (R-Vets Sleep)
Acronym: R-Vets Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-1056
Record Dates: First submitted 2017-11-28; First posted 2017-12-07 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Insomnia; Mental Health Functioning; Physical Health Functioning
Keywords: CBT-I; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized Intervention 1 (Experimental): A web-based program will deliver components of CBT-I on a time and event-based schedule. Pre and Post-Intervention assessments will be administered to determine the efficacy of the intervention.
  Interventions: Behavioral: Computerized Cognitive Behavioral Therapy for Insomnia
- Computerized Intervention 2 (Active Comparator): A web-based program will deliver components of sleep education via an Internet platform. Pre and Post-Intervention assessments will be administered to determine the efficacy of the intervention.
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: Computerized Cognitive Behavioral Therapy for Insomnia — A computerized insomnia intervention that employs the same behavioral, educational, and cognitive treatment components that underlie non-computerized CBT-I.
  Other Names: cCBT-I
  Arms: Computerized Intervention 1
Behavioral: Sleep Education — A web-based program will deliver components of sleep education via an Internet platform
  Arms: Computerized Intervention 2

SUMMARY:
Insomnia is a major problem among veteran populations. Insomnia impacts physical and mental health functioning and is associated with reduced quality of life. Cognitive Behavioral Therapy for Insomnia (CBT-I) is one of the most promising treatments for insomnia; however, access to CBT-I is severely limited by a lack of trained clinicians within the Veterans Health Administration (VHA). There is a critical need to offer innovative approaches to meet the demand and need for insomnia treatment. Leveraging technology to meet treatment demands is consistent with service delivery models based upon stepped care principles. This randomized controlled trial will determine whether a computerized, self-guided, web-based version of CBT-I is efficacious in reducing insomnia symptoms and improving functioning compared to a computerized program control.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 89
2. Eligible to receive care through VA ECHCS
3. Reliable access to the Internet
4. English speaking
5. Able to provide informed consent
6. Current insomnia diagnosis as defined by Diagnostic and Statistical Manual of Mental Disorders 5 (DSM 5) criteria

Exclusion Criteria:

1. Currently enrolled in/participating in other intervention research studies
2. Other untreated sleep disorders (e.g., sleep apnea, periodic limb movement)
3. Currently receiving formal psychological treatment for insomnia (not including sleep medications)
4. Past 3 month change in schedule and/or dosage of medications that are designed to improve/impact sleep
5. History of Bipolar Disorder (with manic episodes), Schizophrenia, Schizoaffective Disorder, or a Psychotic Disorder
6. Untreated seizures or seizure disorder
7. Physical illness that is active, unstable, degenerative, and/or progressive
8. Currently pregnant or plan to become pregnant in the next 6 months
9. Irregular work schedule, shift work, and/or life changes (e.g., new baby) interfering with regular sleep patterns
10. Significant cognitive impairment, as determined by chart review and/or during screening, that would interfere with ability to engage in SHUTi
11. Current non-alcohol Substance Use Disorder, excluding Cannabis Use Disorder, as determined by chart review and/or self-report screen of drug use (> 1 time) in past 3 months
12. Current alcohol use diagnosis, as determined by SCID 5 module, in the past 3 months

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-04-28 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Symptom Severity; Time 1 to Time 2 | Baseline and 9 weeks
  The primary analysis will be the intent-to-treat comparison between groups of the change in insomnia symptom severity as measured by the Insomnia Severity Index (ISI) from Time 1 to Time 2. Statistical inference regarding the difference between intervention groups will be based on the estimated coefficient for a group indicator variable in each of three analysis of covariance models with the change from Time 1 to Time 2 for each outcome serving as the dependent variable. Additional covariates will include the baseline value of the outcome to improve the precision of the estimate, and any potential confounders discovered in the randomization check.
Change in Mental Health; Time 1 to Time 2 | Baseline and 9 weeks
  The primary analysis will be the intent-to-treat comparison between groups of the change in Mental Health summary score, as measured by the Veteran's SF-36, from Time 1 to Time 2. Statistical inference regarding the difference between intervention groups will be based on the estimated coefficient for a group indicator variable in each of three analysis of covariance models with the change from Time 1 to Time 2 for each outcome serving as the dependent variable. Additional covariates will include the baseline value of the outcome to improve the precision of the estimate, and any potential confounders discovered in the randomization check.
Change in Physical Health ; Time 1 to Time 2 | Baseline and 9 weeks
  The primary analysis will be the intent-to-treat comparison between groups of the change in Physical Health summary score, as measured by the Veteran's SF-36, from Time 1 to Time 2. Statistical inference regarding the difference between intervention groups will be based on the estimated coefficient for a group indicator variable in each of three analysis of covariance models with the change from Time 1 to Time 2 for each outcome serving as the dependent variable. Additional covariates will include the baseline value of the outcome to improve the precision of the estimate, and any potential confounders discovered in the randomization check.
Change in Insomnia Symptom Severity; Time 1 to Time 3 | Baseline and 6 Months
  A similar analysis will be performed for the above noted insomnia symptom severity outcome on the change from Time 1 to Time 3 to determine persistence of group differences to six-months post-intervention.
Change in Mental Health; Time 1 to Time 3 | Baseline and 6 Months
  A similar analysis will be performed for the above noted Mental Health summary score, as measured by the Veteran's SF-36, on the change from Time 1 to Time 3 to determine persistence of group differences to six-months post-intervention.
Change in Physical Health; Time 1 to Time 3 | Baseline and 6 Months
  A similar analysis will be performed for the above noted Physical Health summary score, as measured by the Veteran's SF-36, on the change from Time 1 to Time 3 to determine persistence of group differences to six-months post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sarra Nazem, PhD, Principal Investigator — VHAECH
Locations (1):
- Rocky Mountain Regional VA, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No